CLINICAL TRIAL: NCT00868972
Title: Percutaneous Renal Stenting in Renovascular Disease With or Without Distal Atheroembolic Protection
Brief Title: Renal Stenting With Distal Atheroembolic Protection
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Prof. Giancarlo Mansueto, Università di Verona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MOMPF-01
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2010-01-25 (Estimated); Status verified 2010-01

CONDITIONS: Renal Artery Obstruction; Renovascular Hypertension
Keywords: Renal Artery Obstruction; renovascular hypertension; stent; Kidney Failure; embolic protection
MeSH Terms: conditions — Renal Artery Obstruction; Hypertension, Renovascular; Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Embolic protection (Active Comparator): Percutaneous renal stenting using a distal embolic protection device (filter wire ex; Cordis Endovascular, USA).
  Interventions: Procedure: Percutaneous renal stenting intervention; Device: Distal embolic protection
- No embolic protection (Sham Comparator): Percutaneous renal stenting intervention without embolic protection
  Interventions: Procedure: Percutaneous renal stenting intervention

INTERVENTIONS:
Procedure: Percutaneous renal stenting intervention — Percutaneous renal stenting intervention
Device: Distal embolic protection — Distal embolic protection device (filter wire ex; Cordis Endovascular, USA).
  Arms: Embolic protection

SUMMARY:
Atherosclerotic renal artery stenosis (ARAS) is associated with progressive loss of renal function, refractory hypertension and flushing edema, responsible for mortality and morbidity, especially in the elderly. Current treatment includes restoration of the renal arterial lumen by endovascular stent placement and/or intensive medical therapy. There is no unanimous consent on which patients could benefice of the endovascular procedure due to the high rate of renal adverse events especially linked to atheroembolic disease. Recently, renal revascularization using a device which consents distal embolic protection of the kidney demonstrated to be a "safe" auxiliary procedure in a few non randomized studies. Interestingly atheromatous debris was detected in 60 to 80% of these devices analyzed after the procedure suggesting that these devices could prevent atheroembolism in a substantial proportion of patients. On the other hand, only a randomized controlled study can prove that renal stent with distal embolic protection is superior to renal stent alone in preserving kidney function.

Therefore, the present study aims to compare the effects of renal artery stent placement with or without distal embolic protection on renal function in ARAS patients.

Method:

Patients with an ARAS of ≥70% and hypertension not responsive to at least 2 antihypertensive medications and/or renal failure (estimated GFR <60 mL/min/1.73 m2 are randomly assigned to stent placement alone or stent placement with distal embolic protection (FILTER WIRE EX; Cordis Endovascular, USA).

Other medications consist of statins, anti-hypertensive drugs and antiplatelet therapy. Patients are followed for 3 months. The primary outcome of this study is a statistical significant difference in kidney function measured as Cr clearance and cystatin C level in the 2 groups at three months. The trial will include 150 patients.

DETAILED DESCRIPTION:
This is a randomized trial of patients with an ostial ARAS and refractory hypertension and or renal failure. Patients will be randomized to:

(i) renal artery stent placement with distal embolic protection (ii) renal artery stent placement without distal embolic protection To both groups an optimal medical treatment consisting of antihypertensive, lipid-lowering and antiplatelet therapy will be added.

Patients with an ostial ARAS associated with an estimated GFR of <60 mL/min/1.73m2 according to the MDRD formula and/or refractory hypertension are enrolled in this trial. Ostial ARAS is defined as a luminal reduction of ≥70% of the renal artery within 1 cm of the aortic wall, in the presence of atherosclerotic changes of the aorta. Stenosis evaluation can be performed on intra-arterial angiography.

Medical therapy: Irrespective of baseline serum cholesterol values, the patients will be treated with lipid-lowering therapy: 10 mg of rosuvastatin. Any lipid-lowering medication currently used is discontinued and replaced by rosuvastatin. Hypertension is treated with the following drugs: ACE-inhibitors together, loop diuretic, dihydropyridine calcium antagonists. The target BP is <140/90 mmHg. Patients will receive anti-platelet therapy, aspirin 75-100 mg/od plus ticlopidine 250 mg bid for one month. Considering that smoking is a major renal risk factor, smokers will be advised to stop.

Medical therapy is identical in the two treatment arms. In both groups patients will start with aspirin 100 mg/od and ticlopidine 250 mg bid at least five days before admission. The stent (Palmaz-Corinthian IQ/Palmaz Genesis, Johnson & Johnson Medical, NV/SA) will be placed during an in-patient admission according to a standardized protocol. To Patients randomized to the embolic protection the device (FILTER WIRE EX; Cordis Endovascular, USA) will be placed distal to the arterial stenosis before stent placement.

Randomization will be done using random numbers tables The only people aware of the assigned procedure will be the radiologists' team. Researchers and technicians who will follow the patients and analyze the plasma and urinary samples will be blinded to the assigned treatment.

Clinical follow-up is scheduled after 1 and 3 months. Analysis of results: The difference in the mean change of cystatin C respect to baseline between both treatment arms will be assessed including 95% confidence intervals (95% CI). The effects on renal function of the two treatment strategies will be evaluated with multivariate linear regression analysis, considering also the eventual role of age, smoking, diabetes, lipids level, proteinuria, bilateral or unilateral renal artery stenosis, BP and renal function at baseline

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Ostial atherosclerotic renal artery stenosis ≥70% on intra-arterial angiography
* Well documented history of hypertension (>140/90 mmHg) non responsive to the use of 2 or more antihypertensive medications and/or
* Estimated glomerular filtration rate <60 ml/min/1.73m2 according to the MDRD formula, on two occasions within one month

Exclusion Criteria:

* Declined informed consent
* Renal longitudinal diameter < 8 cm
* Any anatomical reasons that make impossible the PTRA and or the positioning of the distal embolic protection device
* Estimated glomerular filtration rate <30 ml/min/1.73m2 according to the MDRD formula or on dialysis
* Allergy to the contrast medium used during angiography
* Other conditions associated with (within 6 months) poor prognosis
* Myocardial infarction, unstable angina or stroke <1 month before planned date of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Differences in renal function loss (measured as Cr clearance and/or cystatin C) after 1 and 3 months of follow-up | 3 months

SECONDARY OUTCOMES:
Acute complications, especially atheroembolism | 3 months
Evaluations of the covariates associated with a better outcome in the atheroembolic device group | 3 months
Blood pressure control (number of medication needed to keep BP<140/90 ) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Mansueto, MD, professor, Principal Investigator — Univerista di Verona
Locations (1):
- Azienda Ospedaliera di Verona, Policlinico G.B. Rossi, Verona, Italy